CLINICAL TRIAL: NCT06546163
Title: The Effects of Heart Rate Variability Biofeedback on College Students With Disordered Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Sunny Wonsun Kim, Ph.D, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00018977
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Eating Disorders; Eating, Binge; Anorexia Nervosa/Bulimia; Eating Disorder Binge; Heart Rate Variability; Psychological Distress; Emotion Regulation; Autonomic Nervous System
Keywords: Psychosocial health; Heart rate variability biofeedback; Eating disorder; College students
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia; Anorexia Nervosa; Binge-Eating Disorder; Emotional Regulation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline and HRVB group (Experimental): In-person baseline surveys (using paper and pen survey) before the random assignment to HRVB arm. This group will receive a standardized HeartMath© Inner balance device and HRV biofeedback training session at the start of the two-week intervention period. They will be asked to attend one-on-one 30-minute HRVB training session and asked to practice their HRV biofeedback skills at home for 10 minutes each day for a two-week period. Participants will receive a weekly email notification and reminder phone call to complete their at-home practice of HRVB.
  Interventions: Behavioral: Baseline survey; Behavioral: Heart rate variability biofeedback
- Baseline and HRVB waitlist (Other): In-person baseline surveys (using paper and pen surveys) before the random assignment to HRVB waitlist group. After the baseline data collection, for two weeks, they will be provided educational material regarding education materials and coping with stress and they will be encouraged to read them during the two weeks. At the end of the two-week period, participants will be scheduled for a final in-person session including T2 survey and HRV assessment. They will be also provided HRVB training session at T2.
  Interventions: Behavioral: Baseline survey; Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Baseline survey — Baseline surveys contains a series of scaled questions, including sociodemographic variable (age, sex, etc), profile of mood states, perceived stress scale, Eating Loss of Control scale, Eating Disorder Examination Questionnaire, Brief Resilience Scale- BRS,Heart Rate Variability and coherence measures
  Other Names: Baseline questionnaire
Behavioral: Heart rate variability biofeedback — Participants randomized to the intervention arm will receive a standardized HRV sensor and accompanying smartphone app, and a 30-minute HRVB training to use the biofeedback signals to generate a resonant frequency pattern of HRV (coherence) after collecting data at baseline in person. Participants will be asked to practice their HRVB skills at home for 10 minutes for two weeks.
  Arms: Baseline and HRVB group
Behavioral: Educational materials — Participants randomized to the waitlist control arm will receive educational materials on eating disorders and stress management and will be sent home with these materials after completing the baseline survey. They will be encouraged to read the materials over the next two weeks before coming in for T2 survey.
  Arms: Baseline and HRVB waitlist

SUMMARY:
The goal of this clinical trial study is to test the heart rate variability biofeedback training in female college students with eating disorders and compare the results between intervention and control group. The main questions it aims to answer are:

* How does heart rate variability biofeedback (HRVB) training impact behaviors related to eating disorders (EDs) and the perceived stress associated with these behaviors?
* What difference are observed in the quality of life and stress responses between individuals trained in HRVB protocol and those in the wait list condition?
* Does HRVB training enhance heart resilience and improve the ability to cope with psychosocial stressors in young women with eating disorders, compared to those in the wait list condition?

Participants will be asked to do the following steps:

* Baseline heart rate variability assessment and completion of the baseline questionnaire
* HRVB training session and two weeks of at-home HRVB practice-10 minutes daily, (intervention group)
* Post-intervention questionnaire completion and heart rate variability assessment
* Optional interview (for intervention group) and HRVB training session (for control group)

Researchers will compare the results of intervention group with control group to see if the participants improve in levels of emotional health, quality of life, and resilience.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aimed at examining the effect of Heart Rate Variability Biofeedback (HRVB) in female college students with eating disorders. The primary objective of the study is to determine whether HRVB can positively impact the psychosocial health and well-being.

Participants are the female college students aged 18 and above. The number of 30 female college students will participate in the study and they will be randomly assigned to either the HRVB intervention group or the control group (15 for each group). Total Duration of the study will be 2 weeks from the time of enrollment to completion.

Participants are required to visit the lab twice - for baseline and final data collection. They undergo initial assessments before any intervention, including a 3- minute baseline HRV assessment (Using the HeartMath Pro Plus device equipped with an ear or finger sensor), and questionnaires about mood states, stress levels, and eating behaviors. The intervention group will receive instructions to practice HRVB and practice it at home for 10 minutes daily over a two-week period, totaling approximately 140 minutes. They will receive a routine calls/texts/email from the research team as a reminder to practice HRVB sessions as well. Final Data Collection will be done at the end of the two-week intervention period for both groups. Participants from the intervention group will have the option to participate in a brief interview to provide feedback on their experiences with the HRVB intervention, and those in control group will receive HRVB training.

All procedure is designed to prioritize participant comfort and privacy, with informed consent being a crucial part of the enrollment process.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as female
* be 18 years of age or older
* be currently enrolled as a college student at ASU
* have experienced or are currently experiencing an eating problem.

Exclusion Criteria:

* have major medical or psychiatric illness
* have conditions that could interfere with HRV data accuracy, such as medications affecting heart rhythm, those with a pacemaker or heart transplant
* use of medications affecting eating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identify as female
Enrollment: 21 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Heart Rate Variability (HRV and coherence scores) at 2 weeks | Baseline (T1), 2 weeks after (T2)
  The Emwave Pro Plus device from HeartMath will be used to collect HRV data and heart rate using a 3-minutes "neutral" protocol (we call "waiting at the bus stop" implying that no particular intent for breath or mindful state is to be evoked) to understand the benefits of HRVB. In addition, HRV measures will be obtained for the 1-minute paced breathing period to understand the effects of paced breathing on HRV. The following precautions will be provided as instructions to participants prior to data collection: no coffee, tea, or caffeinated drinks such as energizing drinks in the 2 hours before the data collection, and no alcohol consumption during 24 hours prior to the data collection.

SECONDARY OUTCOMES:
Changes from Baseline Profile of Mood States (POMS) short version (Psychological Distress) at 2 weeks | Baseline (T1), 2 weeks after (T2)
  Psychological distress will be measured using the Profile of Mood States (POMS) short version (15 items, 5-point Likert scale; 0=not at all, 4=extremely). The POMS is one of the most frequently used and validated scales in studies of psychosocial interventions for cancer patients. The POMS Total Mood Disturbance (TMD) score has been shown to be most sensitive to interventions designed to manage mood or reduce stress. The POMS consists of the TMD dimensions (tension-anxiety; depression-dejection; anger-hostility; and confusion-bewilderment) (Cronbach's a = .93) to be used in the current study as a secondary outcome measure; and two others (fatigue-inertia; vigor-activity) will be documented. Total of Mood Disturbance= (anxious+depression+anger+fatigue)- vigor (Range from 12 to 48). The higher values represent a worse emotional well-being.
Changes from Baseline on Perceived Stress Scale | Baseline (T1), 2 weeks after (T2)
  Perceived stress will be measured using the Perceived Stress Scale (PSS). (10 items, 5-point Likert scale; 0=never, 4=very often). The PSS is one of the most frequently used and validated scales for stress assessment. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. (Cronbach's a = .82) to be used in the current study as a secondary outcome measure. The higher values represent higher perceived stress.
Changes from Baseline on Loss of Control eating brief (LOCES-B) Scale | Baseline (T1), 2 weeks after (T2)
  Loss of control over eating will be measured using LOCES-B. It is a 7-item scale, with a 5-point Likert scale; 1= Never, 5=Always). It is a reliable and valid measure of loss of control over eating. (Cronbach's α = .92). Individual scores on LOCES-B can range between 5- 35 with higher scores indicating greater loss of control over eating. Higher scores on the LOCES-B total score indicate greater body image dissatisfaction, more internalizing symptoms, and lower trait effortful control.
Change from baseline on Eating Disorder Examination Questionnaire | Baseline (T1), 2 weeks after (T2)
  The Eating Disorder Examination Questionnaire (EDE-QS) is a 12-item self-report questionnaire used for the assessment of eating disorder pathology. The EDE-QS has a response scale ranging from 0 to 3 that captures essential symptoms of Anorexia Nervosa, Bulimia Nervosa, and Binge Eating Disorder. The possible range of scores on the scale ranges from 0 to 36 and higher scores indicate greater ED symptoms. ED symptoms are reported for the preceding seven days. Cronbach's alpha obtained in this sample was .91 indicating excellent internal consistency. It is a reliable and valid measure to assess eating disorder pathology.
Change from baseline on Brief Resilience Scale (BRS) | Baseline (T1), 2 weeks after (T2)
  The Brief Resilience Scale is a six-item scale used to measure resilience. The respondents were asked to indicate how well each statement described their behavior and actions on a 5-point Likert-type scale, ranging from "1" = does not describe me at all to "5" = describes me very well. The range of possible scores on BRS is from 6-30. There are three positively worded items and three negatively worded items. The three negative items will be reverse-coded during scoring It is a valid and reliable measure of resilience. (Cronbach's α = .85).

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States